CLINICAL TRIAL: NCT05926388
Title: The Effect of Video-Assisted Instruction in Type 2 Diabetes Patients' Insulin Self-Management and Insulin Administration Skills
Brief Title: Video-Assisted Instruction in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Elif Günay İsmailoğlu, Associate Professor, Izmir Bakircay University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BU-SBF-EI-001
Record Dates: First submitted 2023-06-02; First posted 2023-07-03 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Education, Patient
Keywords: self-management; Type 2 diabetes mellitus; video-assisted instruction
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video-assisted training group (Experimental): The researcher will train the patients with video-assisted on insulin therapy and administration.
  Interventions: Other: Video-assisted training

INTERVENTIONS:
Other: Video-assisted training — Patients will be given training on insulin therapy and management using lecture, question-answer, video and demonstration methods.

SUMMARY:
The aim of the study of examine the effect of video-assisted instruction on Type 2 diabetes patients' insulin treatment self-management and insulin administration skills. The research will be conducted as a single group pre-test post-test quasi-experimental study. The sample of the study will be consisted of 50 patients with Type 2 Diabetes. Before the training, the patients will be self-injected a dose of insulin. After giving verbal training, the patients will watch a video recording of insulin treatment and administration. The author will be evaluated the patients' insulin treatment self-management and insulin administration skills after the training.

DETAILED DESCRIPTION:
The aim of the study of examine the effect of video-assisted instruction on Type 2 diabetes patients' insulin treatment self-management and insulin administration skills. The research will be conducted as a single group pre-test post-test quasi-experimental study. The sample of the study will be consisted of 50 patients with Type 2 Diabetes. Before the training, the patients will be self-injected a dose of insulin. After giving verbal training, the patients will watch a video recording of insulin treatment and administration. The author will be evaluated the patients' insulin treatment self-management and insulin administration skills after the training.

ELIGIBILITY:
Inclusion Criteria

* 18-65 years
* No hearing or communication problems
* Self-injecting insulin

Exclusion Criteria

* Health care professionals
* Chronic complications
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Insulin Treatment Self-Management Scale 1 (Questionnaire) | Seven days after the training
  Patients' self-injection practices will be evaluated.
Insulin Treatment Self-Management Scale 2 (Questionnaire) | Five weeks after the training
  Patients' self-injection practices will be evaluated.
Insulin Administration Observation Form 1 | Seven days after the training
  The scale identifies knowledge and skill levels of patients.
Insulin Administration Observation Form 2 | Five weeks after the training
  The scale identifies knowledge and skill levels of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- izmir Bakircay University, Izmir, Menemen, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No